CLINICAL TRIAL: NCT04128137
Title: Evaluation of Efficacy and Tolerance of Fludrocortisone (Flucortac) in the Treatment of Orthostatic Neurogenic Hypotension
Brief Title: Efficacy and Tolerance of Flucortac in Patients With Orthostatic Neurogenic Hypotension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: H.A.C. PHARMA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-003905-25
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Neurogenic Orthostatic Hypotension
MeSH Terms: interventions — Fludrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fludrocortisone (Experimental): FLUCORTAC® 50 μg (tablet breackable). One tablet during the first week. Then 2 tablets during the second week. Then 3 tablets during the third week and finally 4 tablets during the 4th week. Maximum of 200μg/day.
  Interventions: Drug: Fludrocortisone
- Placebo (Placebo Comparator): placebo of flucortac and same diagram of administration
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fludrocortisone — 50 µg/day during one week then augmentation of 50 µg each weeks until a maximum dose of 200 µg/day. And a maintenance phase of 4 weeks at a stable dose
  Other Names: Flucortac
  Arms: fludrocortisone
Other: Placebo — 50 µg/day during one week then augmentation of 50 µg each weeks until a maximum dose of 200 µg/day. And a maintenance phase of 4 weeks at a stable dose
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of a 4-week fludrocortisone (FLU) treatment on systolic blood pressure depression after 5 minutes of active orthostatism in patients with neurogenic orthostatic hypotension (HON) symptomatic, despite treatment with non-drug measures with or without midodrine.

DETAILED DESCRIPTION:
The objective of the study is to demonstrate the efficacy of FLU on systolic blood pressure depression in patients with neurogenic orthostatic hypotension. The study is randomised versus placebo.Each patient will be followed for a maximum of 5 months, with no more than 8 visits to the investigator (V0 at Day-7, V1 at D0, V2 at D7, V3 at D+14, V4 at D+21, V5 at D+ 28, V6 at D+56 and V7 only for patients on the FLU arm at D+140.

The presence of a comparator control group with placebo permits to evaluate the efficacy and the tolerance of FLU independently of the natural evolution of the pathology, in patients benefiting from a non-drug or possibly medicated treatment (midodrine) but insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of orthostatic hypotension (HO), ie a blood pressure drop> 20 and / or 10 mmHg within 3 minutes after active and symptomatic lifting
* Patient suffering from a neurological disease
* orthostatic neurogenic hypotension persistent and symptomatic despite non-drug measures

Exclusion Criteria:

* Hypersensitivity to FLU or any of its excipients
* non orthostatic neurogenic hypotension
* History of proven heart failure
* History of left ventricular systolic dysfunction
* Uncompensated hypokalemia
* Patient with poorly balanced Grade 3 hypertension
* Pregnant patient at the time of inclusion
* Nursing patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Systolic BP diminution | 8 weeks
  Systolic BP diminution when moving from supine to standing, measured with a semi-automatic blood pressure monitor
  - AP in upright position: the lowest value of the measurements obtained every minute, for 5 minutes after rising.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel SENARD, MD, Principal Investigator — National Coordinator
Locations (1):
- Hôpital Broca (AP-HP), Paris, France